CLINICAL TRIAL: NCT04022681
Title: Long-term Follow Up of Patients in the Birmingham and Lambeth Liver Evaluation Strategies (BALLETS) Study
Status: Completed | Type: Observational
Sponsor: University of Warwick (Other)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Principal Investigator, Professor Richard Lilford, Professor of Public Health, University of Warwick
Other Study IDs: BALLETS-LT-Followup
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Fatty Liver; Liver Diseases
MeSH Terms: conditions — Fatty Liver; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-specific liver disease: Patients who were categorised as having a non-specific liver disease in the original BALLETS study.
  Interventions: Other: BALLETS

INTERVENTIONS:
Other: BALLETS — Cohort were not exposed to any intervention. There information will be analysed from database searches.

SUMMARY:
This study will follow-up a cohort of patients from the Birmingham and Lambeth Liver Evaluation Strategies (BALLETS) study using a database search based on their individual National Health Service (NHS) numbers. The investigators will interrogate the Hospital Episode Statistics database and the Office of National Statistics database, and examine three categories of end points: death, inpatient attendance primarily due to liver disease, and outpatient attendance primarily due to liver disease.

A logistic regression analysis will then be conducted to determine associations between these end points and the presence, and degree, of fatty liver in the original BALLETS study, adjusted for age, sex, alcohol intake, BMI, and baseline ALT measurement.

DETAILED DESCRIPTION:
The Birmingham and Lambeth Liver Evaluation Strategies (BALLETS) study was a prospective study of people in General Practice who had an abnormal liver function test result. Recruitment took place between 2005 and 2008, and patients were able to be grouped into four primary categories: hepato-cellular disease, hepato-biliary disease, tumour, non-specific with or without fatty liver. This study will focus on the fourth, non-specific, group of which there were 1,237 patients.

This study will follow-up this cohort of patients using a database search based on their individual National Health Service (NHS) numbers. The investigators will interrogate the Hospital Episode Statistics database (health outcomes) and the Office of National Statistics database (death), and examine three categories of end points: death, inpatient attendance primarily due to liver disease, and outpatient attendance primarily due to liver disease. Deaths would be sub-categorised as including liver disease, or not.

A logistic regression analysis will then be conducted to determine associations between these end points and the presence, and degree, of fatty liver in the original BALLETS study, with adjustment for age and sex. Similar age- and sex-adjusted analyses will be conducted to investigate the association with other patient risk factors - alcohol intake and BMI. The analyses will be repeated incorporating an additional adjustment for baseline Alanine Aminotransferase (ALT) measurement.

ELIGIBILITY:
Inclusion Criteria:

* Adult with abnormal liver function test (LFT) result

Exclusion Criteria:

* Pre-existing or obvious liver disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in primary care with no known liver disease, who had a liver function test (LFT)
Sampling Method: Non-Probability Sample
Enrollment: 1237 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients who Died | From date of recruitment until the date of death, up to 14 years
  Death of patient, sub-categorised as either including liver disease, or liver disease not mentioned

SECONDARY OUTCOMES:
Number of patients attending inpatient department, primary reason liver disease | From date of recruitment until the date of database search, up to 14 years
  Number of patients attending hospital inpatient department, with their primary reason for attendance being liver disease, as measured by the hospital episode statistics database.
Number of patients attending outpatient department, primary reason liver disease | From date of recruitment until the date of database search, up to 14 years
  Number of patients attending hospital outpatient department, with their primary reason for attendance being liver disease, as measured by the hospital episode statistics database.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Lilford, FMedSci, Principal Investigator — University of Warwick

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not available to be shared.

REFERENCES:
- [Background] Lilford RJ, Bentham L, Girling A, Litchfield I, Lancashire R, Armstrong D, Jones R, Marteau T, Neuberger J, Gill P, Cramb R, Olliff S, Arnold D, Khan K, Armstrong MJ, Houlihan DD, Newsome PN, Chilton PJ, Moons K, Altman D. Birmingham and Lambeth Liver Evaluation Testing Strategies (BALLETS): a prospective cohort study. Health Technol Assess. 2013 Jul;17(28):i-xiv, 1-307. doi: 10.3310/hta17280. PMID 23834998